CLINICAL TRIAL: NCT05773391
Title: A Prospective Phase II Study About Mechanism Exploration of Anti-HER-2 Small-molecule Tyrosine Kinase Inhibitor-related Diarrhea and Establishment of Prevention and Treatment Model in HER2+ Breast Cancer
Brief Title: Mechanism Exploration of Anti-HER-2 Small-molecule Tyrosine Kinase Inhibitor-related Diarrhea and Establishment of Prevention and Treatment Model(Measure)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Chief Physician, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-2022-01
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diarrhea group (Experimental): Patients with diarrhea after taking pyrrolidine/naratinib，implement intervention (Yihuo 0.2g po bid+ Gold bifidum 2g po tid)
  Interventions: Drug: Take probiotics
- No diarrhea group (No Intervention): Patients without diarrhea after taking pyrrolidine/naratinib

INTERVENTIONS:
Drug: Take probiotics — Take medication for 21 days (Yihuo 0.2g bid+ Jin Bifid2g tid)
  Arms: Diarrhea group

SUMMARY:
Small-molecule tyrosine kinase inhibitors (TKI) that target HER2 are routinely used to treat patients with HER2 (+) breast cancer. The main adverse reactions included diarrhea, nausea, and rash, among which diarrhea had the highest incidence. It can reduce the quality of life and medication compliance of patients, and further affect the efficacy of TKI anti-tumor therapy. Therefore, the investigators conducted this study to establish a risk assessment model before TKI treatment, in order to screen out the high-risk population and influencing factors of TKI-associated diarrhea, and planned to carry out corresponding animal experiments to verify the relationship between various mechanisms and the main mechanism in TKI-associated diarrhea and to explore the corresponding treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* Plan to take pyrrolidine or naratinib for ≥ 28 days;
* HER2 positive female patients with breast cancer aged ≥ 18 years and ≤ 65 years;
* Patients with the following treatment schemes: 1. Pirotinib/naratinib monotherapy 2. Pirotinib/naratinib combined endocrine therapy; 4. The ECOG score is 0-1;
* Life expectancy ≥ 6 months;
* Patients who followed diet intervention after enrollment;
* Volunteer to join the study, sign the informed consent form, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

* People who may be allergic to pyrrolidine, naratinib or excipients;
* There are many factors that affect the absorption of oral drugs, such as inability to swallow, nausea and vomiting;
* Patients with biliary obstruction;
* Participate in other clinical trials related to diarrhea;
* Pregnant and lactating women, women with fertility and positive baseline pregnancy test, or women of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period;
* According to the judgment of the investigator, there are concomitant diseases (including but not limited to severe hypertension and severe diabetes beyond drug control) that seriously endanger the patient's safety or affect the patient's completion of the study;
* Have taken other drugs that may cause diarrhea adverse reactions within 3 weeks before enrollment;
* There are drugs with high probability of causing diarrhea adverse reactions in patients' combined medication;
* Any other situation in which the researcher believes that the patient is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-12 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Diarrhea grading | 28 days
  Score according to the diarrhea grading：grading score： 0（None）；1（Increased bowel movements < 4 times per day compared to before treatment）； 2（Increased bowel movements 4 to 6 times/day or night compared to before treatment）；3（ Increased number of stools ≥ 7 times/day compared with before treatment, fecal incontinence, severe abdominal pain or fecal incontinence, affecting daily activities and requiring hospitalization）； 4（life-threatening (e.g. circulatory failure））；5（Death）.

SECONDARY OUTCOMES:
Time of the first occurrence of diarrhea | 28 days
  The median time of the first occurrence of diarrhea
Duration of diarrhea | 28 days
  The median duration of diarrhea
Time of the first occurrence of grade 3 diarrhea | 28 days
  The median time of the first occurrence of grade 3 diarrhea
Duration of grade 3 diarrhea | 28 days
  The median duration of grade 3 diarrhea
Adverse events | 28 days
  Occurrence of other adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China